CLINICAL TRIAL: NCT06108882
Title: Effects of Manual Ischemic Compression With and Without Strain Counter Strain Technique on Sternocleidomastoid Tightness With Forward Head Posture
Brief Title: Effects of Manual IC With and Without SCS on SCM Tightness With FHP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0147
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Neck Pain
Keywords: Disability; Forward head posture; Pain; ROM; Sternocleidomastoid
MeSH Terms: conditions — Neck Pain; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual Ischemic Compression with Strain Counter Strain technique (Experimental): Participants in this group will receive Manual Ischemic Compression with Strain Counter Strain technique.
  Interventions: Other: Experimental: Manual Ischemic Compression with Strain Counter Strain technique
- Manual Ischemic Compression (Active Comparator): Participants in this group will receive only Manual Ischemic Compression
  Interventions: Other: Active Comparator: Manual Ischemic Compression

INTERVENTIONS:
Other: Experimental: Manual Ischemic Compression with Strain Counter Strain technique — The duration of intervention will be 6 weeks, 3 sessions a week, a total of 18 sessions will be given to the study participants. Each session will last for 30 to 45 minutes.
  Arms: Manual Ischemic Compression with Strain Counter Strain technique
Other: Active Comparator: Manual Ischemic Compression — The duration of intervention will be 6 weeks, 3 sessions a week, a total of 18 sessions will be given to the study participants. Each session will last for 30 to 45 minutes.
  Arms: Manual Ischemic Compression

SUMMARY:
The aim of this study is to compare the effects of Manual Ischemic Compression with and without Strain Counterstrain technique on CVA, ROM, pain and disability among FHP individuals with SCM tightness.

DETAILED DESCRIPTION:
Forward head posture is defined by excessive extension at upper cervical spine(C1-C3) and flexion at lower cervical spine (C4-C7) that increases cranial rotation angle and decreases craniovertebral angle (CVA) because of the altered relative position of the head with respect to the line of gravity. The bubble inclinometer is a gravity-based tool used to measure the cervical range of motion and to assess SCM muscle length. FHP also leads to muscles imbalance and SCM tightness as well. The Numerical Pain Rating Scale (NPRS) are most frequently used to quantify pain intensity and NDI for neck disability.

A RCT study compare the effects of IC and SCS in patients with upper trapezius trigger points. For four weeks, the therapy was given three days a week. As an outcome indicator, the NPRS, NDI, and cervical lateral flexion were used. The outcome measures were evaluated at baseline, after the second week, and after the fourth week: The ischemic compression and strain counterstrain intervention, which lasted for four weeks, significantly improved cervical range of motion, reduced pain intensity, and reduced cervical disability. However, the intergroup comparison revealed that both interventions were equally effective, and none of them outperformed the others.

Most of the studies compared digital ischemic compression as a common treatment with dry needling or other soft tissue mobilizations specially to treat trapezius trigger points but there are few studies specifically investigating comparative effects of Manual Ischemic Compression with and without Strain Counterstrain for management purpose of muscle tightness in individuals with FHP. While various treatment options exist for FHP, limited research directly compares the comparative outcomes of Strain Counterstrain and Ischemic Compression techniques. Due to lack of comparative evidence regarding the efficacy of these specific interventions, there is a need to bridge this gap by investigating and comparing the effectiveness of these interventions by using highly reliable and valid outcome measures in order to provide healthcare professionals and individuals with evidence-based guidance for optimal FHP management and SCM tightness.

ELIGIBILITY:
Inclusion Criteria:

* Neck pain (Numeric Pain Rating Scale >3)
* Craniovertebral angle (CVA) less than 51
* Shortened SCM muscle

Exclusion Criteria:

* Neck pain with whiplash or headache, neurological disorder
* History of previous head, neck, cervical spine or shoulder surgery
* Infection or inflammatory arthritis in the cervical spine
* History of cervical radiculopathy

  * Diagnosed fibromyalgia and myopathy
  * History of cancer

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-05-08 (Actual); Primary Completion 2023-12-08 (Estimated); Study Completion 2024-01-08 (Estimated)

PRIMARY OUTCOMES:
Numeric pain rating scale (NPRS) | 6 weeks
  Changes from baseline Numeric pain rating scale is The 11-point scale used to capture the patient's level of pain. The scale is anchored on the left with the phrase ''no pain'' and on the right with the phrase ''worst imaginable pain.'' Patients rate their current level of pain and their worst and least amount of pain in the last 24 hours.
Neck disability index (NDI) | 6 weeks
  Changes from baseline the NDI is a self-report questionnaire with 10 items: Pain intensity, personal care, lifting, work, headaches, concentration, sleeping, driving, reading and recreation. The response to each item is rated on a six-point scale from 0 (no disability) to 5 (complete disability). The numeric responses for each item are summed for a total score ranging between 0 and 50; however, some evaluators have chosen to multiply the raw score by 2 and then report the NDI on a 0-100% scale. Higher scores represent increased levels of related disability among the participants The maximum score is 50. In which 0 to 4 indicates no disability 5 to 14 = mild, 15 to 24 = moderate, 25 to 34 = severe and Above 34 = complete disability(57).
The bubble inclinometer | 6 weeks
  Changes from baseline bubble inclinometer is a gravity-based tool used to measure the cervical range of motion and to assess SCM muscle length based on Kendall's description of muscle length testing principles in which the therapist maximally lengthens the muscle from origin to insertion by stabilizing one end, then slowly elongate the muscle, and then assess the end feel.
Craniovertebral angle (CVA) | 6 weeks
  Changes from baseline To assess the head position of the subjects, the craniovertebral angle (CVA) was measured. The craniovertebral angle is identified as the intersection of a horizontal line passing through the C7 spinous process and a line joining the midpoint of the tragus of the ear to the skin overlying the C7 spinous process. CVA angle less than 51 is considered as FHP.
Modified goniometer | 6 weeks
  Changes from baseline the measurement of craniovertebral angle is from C7 spinous process to tragus of ear by modified goniometer. The craniovertebral angle can be assessed by using modified goniometer to get an accurate estimation of head posture. The modified goniometer was constructed by attaching a perpendicular rod at the fulcrum of half circle universal goniometer, posteriorly. .
Neck ROM | 6 weeks
  Changes from baseline, neck ROM will be taken with the help of goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: Saba Rafique, Masters, Principal Investigator — Riphah International University
Locations (1):
- Amina Physiotherapy and Rehab Center, Nusrat Rashid Medical Complex, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kang NY, Im SC, Kim K. Effects of a combination of scapular stabilization and thoracic extension exercises for office workers with forward head posture on the craniovertebral angle, respiration, pain, and disability: A randomized-controlled trial. Turk J Phys Med Rehabil. 2021 Sep 1;67(3):291-299. doi: 10.5606/tftrd.2021.6397. eCollection 2021 Sep. PMID 34870115
- [Background] Khan A, Khan Z, Bhati P, Hussain ME. Influence of Forward Head Posture on Cervicocephalic Kinesthesia and Electromyographic Activity of Neck Musculature in Asymptomatic Individuals. J Chiropr Med. 2020 Dec;19(4):230-240. doi: 10.1016/j.jcm.2020.07.002. Epub 2020 Nov 24. PMID 33536860
- [Background] Mahmoud NF, Hassan KA, Abdelmajeed SF, Moustafa IM, Silva AG. The Relationship Between Forward Head Posture and Neck Pain: a Systematic Review and Meta-Analysis. Curr Rev Musculoskelet Med. 2019 Dec;12(4):562-577. doi: 10.1007/s12178-019-09594-y. PMID 31773477
- [Background] Sikka I, Chawla C, Seth S, Alghadir AH, Khan M. Effects of Deep Cervical Flexor Training on Forward Head Posture, Neck Pain, and Functional Status in Adolescents Using Computer Regularly. Biomed Res Int. 2020 Oct 5;2020:8327565. doi: 10.1155/2020/8327565. eCollection 2020. PMID 33083487
- [Background] Shiravi S, Letafatkar A, Bertozzi L, Pillastrini P, Khaleghi Tazji M. Efficacy of Abdominal Control Feedback and Scapula Stabilization Exercises in Participants With Forward Head, Round Shoulder Postures and Neck Movement Impairment. Sports Health. 2019 May/Jun;11(3):272-279. doi: 10.1177/1941738119835223. Epub 2019 Apr 23. PMID 31013190
- [Background] Chu ECP, Lo FS, Bhaumik A. Plausible impact of forward head posture on upper cervical spine stability. J Family Med Prim Care. 2020 May 31;9(5):2517-2520. doi: 10.4103/jfmpc.jfmpc_95_20. eCollection 2020 May. PMID 32754534
- [Background] Mylonas K, Angelopoulos P, Billis E, Tsepis E, Fousekis K. Combining targeted instrument-assisted soft tissue mobilization applications and neuromuscular exercises can correct forward head posture and improve the functionality of patients with mechanical neck pain: a randomized control study. BMC Musculoskelet Disord. 2021 Feb 21;22(1):212. doi: 10.1186/s12891-021-04080-4. PMID 33612123
- [Background] Balthillaya GM, Parsekar SS, Gangavelli R, Prabhu N, Bhat SN, Rao BK. Effectiveness of posture-correction interventions for mechanical neck pain and posture among people with forward head posture: protocol for a systematic review. BMJ Open. 2022 Mar 9;12(3):e054691. doi: 10.1136/bmjopen-2021-054691. PMID 35264350
- [Background] Ghamkhar L, Kahlaee AH. Is forward head posture relevant to cervical muscles performance and neck pain? A case-control study. Braz J Phys Ther. 2019 Jul-Aug;23(4):346-354. doi: 10.1016/j.bjpt.2018.08.007. Epub 2018 Aug 22. PMID 30145129
- [Background] Ghan GM, Babu VS. Immediate Effect of Cervico-thoracic Mobilization on Deep Neck Flexors Strength in Individuals with Forward Head Posture: A Randomized Controlled Trial. J Man Manip Ther. 2021 Jun;29(3):147-157. doi: 10.1080/10669817.2020.1834321. Epub 2020 Oct 22. PMID 33090945
- [Background] Chang MC, Choo YJ, Hong K, Boudier-Reveret M, Yang S. Treatment of Upper Crossed Syndrome: A Narrative Systematic Review. Healthcare (Basel). 2023 Aug 17;11(16):2328. doi: 10.3390/healthcare11162328. PMID 37628525
- [Background] Cho J, Lee E, Lee S. Upper cervical and upper thoracic spine mobilization versus deep cervical flexors exercise in individuals with forward head posture: A randomized clinical trial investigating their effectiveness. J Back Musculoskelet Rehabil. 2019;32(4):595-602. doi: 10.3233/BMR-181228. PMID 30584118
- [Background] Alowa Z, Elsayed W. The impact of forward head posture on the electromyographic activity of the spinal muscles. J Taibah Univ Med Sci. 2020 Dec 16;16(2):224-230. doi: 10.1016/j.jtumed.2020.10.021. eCollection 2021 Apr. PMID 33897327
- [Background] Cibulka MT, Herren J, Kilian A, Smith S, Mahmutovic F, Dolles C. The reliability of assessing sternocleidomastoid muscle length and strength in adults with and without mild neck pain. Physiother Theory Pract. 2017 Apr;33(4):323-330. doi: 10.1080/09593985.2017.1302539. Epub 2017 Apr 5. PMID 28379051
- [Background] Young IA PT, DSc, Dunning J PT, DPT, Butts R PT, PhD, Mourad F PT, DPT, Cleland JA PT, PhD. Reliability, construct validity, and responsiveness of the neck disability index and numeric pain rating scale in patients with mechanical neck pain without upper extremity symptoms. Physiother Theory Pract. 2019 Dec;35(12):1328-1335. doi: 10.1080/09593985.2018.1471763. Epub 2018 Jun 1. PMID 29856244
- [Background] Young IA, Dunning J, Butts R, Cleland JA, Fernandez-de-Las-Penas C. Psychometric properties of the Numeric Pain Rating Scale and Neck Disability Index in patients with cervicogenic headache. Cephalalgia. 2019 Jan;39(1):44-51. doi: 10.1177/0333102418772584. Epub 2018 Apr 19. PMID 29673262
- [Background] Joshi R, Poojary N. The Effect of Muscle Energy Technique and Posture Correction Exercises on Pain and Function in Patients with Non-specific Chronic Neck Pain Having Forward Head Posture-a Randomized Controlled Trail. Int J Ther Massage Bodywork. 2022 Jun 1;15(2):14-21. doi: 10.3822/ijtmb.v15i2.673. eCollection 2022 Jun. PMID 35686175
- [Background] Nasb M, Qun X, Ruckmal Withanage C, Lingfeng X, Hong C. Dry Cupping, Ischemic Compression, or Their Combination for the Treatment of Trigger Points: A Pilot Randomized Trial. J Altern Complement Med. 2020 Jan;26(1):44-50. doi: 10.1089/acm.2019.0231. Epub 2019 Oct 3. PMID 31580695
- [Background] Hasuo H, Hashimoto K, Iwamoto H, Miwa N, Kawashima T, Oda A, Sekimoto G. Effect of ischemic compression performed by family caregivers on myofascial pain syndrome and the care burden of the families of patients: a multicenter open-label randomized comparative study. Ann Palliat Med. 2022 Apr;11(4):1179-1190. doi: 10.21037/apm-21-2276. Epub 2021 Dec 6. PMID 34894707
- [Background] Otadi K, Sarafraz H, Jalaie S, Rasouli O. Combining Patient Education With Dry Needling and Ischemic Compression for Treating Myofascial Trigger Points in Office Workers With Neck Pain: A Single-Blinded, Randomized Trial. J Chiropr Med. 2020 Dec;19(4):222-229. doi: 10.1016/j.jcm.2020.02.005. Epub 2020 Nov 24. PMID 33536859
- [Background] Fritz K, Krupa KN, Sina RE, Carr Jr CL. Physiology, Counterstrain and Facilitated Positional Release (FPR). 2023 Nov 13. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK562152/ PMID 32965823
- [Background] Bazzi MO, Sergent SR. Osteopathic Manipulative Treatment: Counterstrain Procedure - Cervical Vertebrae. 2023 Jul 25. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK560846/ PMID 32809681
- [Background] Azam I, Chahal A, Kapoor G, Chaudhuri P, Alghadir AH, Khan M, Kashoo FZ, Esht V, Alshehri MM, Shaphe MA, Khan AR, Singh G. Effects of a program consisting of strain/counterstrain technique, phonophoresis, heat therapy, and stretching in patients with temporomandibular joint dysfunction: [corrected]. Medicine (Baltimore). 2023 Aug 11;102(32):e34569. doi: 10.1097/MD.0000000000034569. PMID 37565891
- [Background] El-Khateeb YS, Mahmoud AG, Mohamed MH, Abd El-Azeim AS. Influence of adding strain-counterstrain to standard therapy on axioscapular muscles amplitude and fatigue in mechanical neck pain: a single-blind, randomized trial. Eur J Phys Rehabil Med. 2022 Aug;58(4):621-629. doi: 10.23736/S1973-9087.22.07194-5. Epub 2022 Jun 6. PMID 35666489
- [Background] Modarresi S, Lukacs MJ, Ghodrati M, Salim S, MacDermid JC, Walton DM; CATWAD Consortium Group. A Systematic Review and Synthesis of Psychometric Properties of the Numeric Pain Rating Scale and the Visual Analog Scale for Use in People With Neck Pain. Clin J Pain. 2021 Oct 26;38(2):132-148. doi: 10.1097/AJP.0000000000000999. PMID 34699406
- [Background] da Silva AC, De Noronha M, Liberatori-Junior RM, Aily JB, Goncalves GH, Arrais-Lima C, de Araujo Vieira LMSM, Mattiello SM. The Effectiveness of Ischemic Compression Technique on Pain and Function in Individuals With Shoulder Pain: A Systematic Review. J Manipulative Physiol Ther. 2020 Mar-Apr;43(3):234-246. doi: 10.1016/j.jmpt.2019.10.013. Epub 2020 Aug 1. PMID 32747150
- [Background] Togha M, Bahrpeyma F, Jafari M, Nasiri A. A sonographic comparison of the effect of dry needling and ischemic compression on the active trigger point of the sternocleidomastoid muscle associated with cervicogenic headache: A randomized trial. J Back Musculoskelet Rehabil. 2020;33(5):749-759. doi: 10.3233/BMR-171077. PMID 31815684
- [Background] Kim SY, An CM, Cha YS, Kim DH. Effects of sling-based manual therapy on cervicothoracic junction in patients with neck pain and forward head posture: A randomized clinical trial. J Bodyw Mov Ther. 2021 Jul;27:447-454. doi: 10.1016/j.jbmt.2021.03.007. Epub 2021 Mar 19. PMID 34391270